CLINICAL TRIAL: NCT01425645
Title: Families Defeating Diabetes: Canadian Intervention for Family-Centered Diabetes Prevention Following Gestational Diabetes (GDM)
Brief Title: Families Defeating Diabetes
Acronym: FDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ruth McManus, MD, FRCPC, Cert Endo, Professor of Medicine, UWO, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RXX
Record Dates: First submitted 2011-08-27; First posted 2011-08-30 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Prevention
Keywords: gestational diabetes; GDM; prevention
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle and behavioural change support (Active Comparator): Interventional arm will be offered a 12 month lifestyle program translating DM prevention issues to the family milieu
  Interventions: Other: FDD program
- control (No Intervention): Control arm will receive standard diabetes prevention care as outlined in the current Canadian diabetes association Clinical Practice Guidelines.

INTERVENTIONS:
Other: FDD program — FDD is a 12 month lifestyle intervention and behavioural support program delivered in the context of the surrounding family
  Arms: Lifestyle and behavioural change support

SUMMARY:
No evidence-based, evaluated, population-appropriate resources exist to translate Type 2 diabetes (T2DM) primary prevention messages to Canadians. Significant barriers to such large-scale interventions include:

* the need to identify, then target specific at-risk populations
* significant time-delays before any program effects on T2DM incidence may manifest.

However, women with gestational diabetes (GDM) are a readily identifiable study cohort at significant risk for recurrent GDM and T2DM-hence GDM women provide important opportunities for rigorous, timely diabetes prevention intervention studies. The investigators propose FDD (Families Defeating Diabetes), a Canadian diabetes prevention intervention uniquely targeting women with recent GDM in the context of their families.

FDD is a 12 month, randomized, controlled T2DM prevention intervention targeting women with recent GDM, within their family context. Five Canadian sites and 177 women will participate. Multifaceted information and behavioural change support will be provided for diet, weight loss, and activity through: seminar, walking groups, electronic updates, password-protected social networking site.

Subjects and controls will be compared for: DM prevention knowledge; diet/activity choices; HbA1C; body habitus at study onset/during study/12 months/24 months.

Consenting immediate family members will have protective knowledge/diet/exercise choices/body habitus measures documented at study onset/12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-50 with recent GDM
* able to speak and write English
* overweight (BMI >25 before pregnancy)
* significant other family members

Exclusion Criteria:

* women with Types 1 or 2 diabetes
* women with BMI under 25

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2012-01; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of study subjects achieving a 7% weight loss | one year post-partum
  Weight loss in intervnetional vs control women will be documented by one year post-partum

CONTACTS AND LOCATIONS:
Locations (1):
- St Josephs Health Care, London, Ontario, Canada